CLINICAL TRIAL: NCT07244315
Title: Cervical Cancer Screening of Postmenopausal Women in Low- and Middle-income Countries Using HPV Self-sampling and Triage by Genotyping and Cytology
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Patrick Petignat, Head of the Gynecologic Division, University Hospital, Geneva
Other Study IDs: N°/537/29/05/2024/CE/CRERSH-OU; AO_2024-00066 (Other: Cantonal Research Ethics Commission of Geneva (CCER, Switzerland))
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Screening; HPV Infections; Cervical Intraepithelial Neoplasia
Keywords: cytology; post-menopausal women; cervical cancer screening
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia | interventions — Papanicolaou Test; Human Papillomavirus DNA Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women from the general population aged 50-65 years old: Women from the general population aged 50-65 years old eligible for screening in the West region of Cameroon.
  Inclusion criteria
  * Women aged 50 to 65 years old;
  * Ability to understand study procedures and accepting voluntarily to participate by signing an informed consent form (ICF).
  Exclusion criteria
  * Women who is pregnant;
  * Women with a condition that interfere with visualization of the cervix;
  * Women with vaginal bleeding outside the menstrual period;
  * Women who have had a total hysterectomy;
  * Women with a history of cervical cancer;
  * Women screened for cervical cancer in the last 5 years or in the last 3 years if HIV-positive;
  * Women in the terminal phase of an illness.
  Interventions: Diagnostic Test: Vaginal specimens for HPV test will be collected by participants themselves using flocked swabs after explanations by co-investigators.

INTERVENTIONS:
Diagnostic Test: Vaginal specimens for HPV test will be collected by participants themselves using flocked swabs after explanations by co-investigators. — Women will perform a self-collected vaginal sample for the detection of high-risk human papillomavirus (HPV) DNA using a molecular assay (HPV DNA test). The sample will be collected using a sterile flocked swab and placed in a transport medium. Laboratory analysis will be conducted at the Mifi District Hospital using the GeneXpert HPV assay (Cepheid, USA).
  Women who test positive for high-risk HPV will undergo cytology triage (Pap test) and, if cytology is positive (≥ASC-US), will be offered thermal ablation at Bafoussam Regional Hospital.
  Other Names: VIA/VILI; Pap smear; Cervical biopsy; Endo-cervical brushing; HPV test

SUMMARY:
Cervical cancer remains a major cause of mortality in low- and middle-income countries, especially among women aged 50 years and older who are often under-screened. In post-menopausal women, the transformation zone is frequently not visible, which makes visual inspection with acetic acid (VIA) less reliable and limits access to adequate screening. Human papillomavirus (HPV) self-sampling offers a simple and acceptable primary screening method, but effective triage options for HPV-positive women in this age group remain limited.

This study aims to evaluate the feasibility and diagnostic performance of a screening strategy based on HPV self-sampling followed by Pap cytology triage among HPV-positive women aged 50 to 65 years in Cameroon. Approximately 500 women will be invited to perform self-HPV testing at the Mifi District Hospital. HPV-positive women will undergo Pap cytology, endocervical brushing and digital cervicography, and eligible participants will receive treatment with thermal ablation at Bafoussam Regional Hospital. Follow-up at 12 months will include repeat HPV testing, cytology, and endocervical brushing.

The primary outcome is the diagnostic accuracy of HPV + cytology triage for detecting CIN2+. Secondary outcomes include prevalence of high-risk HPV, treatment outcomes, acceptability, and adherence to follow-up.

DETAILED DESCRIPTION:
Cervical cancer remains a leading cause of cancer-related mortality among women in low- and middle-income countries (LMICs), including Cameroon. Although most screening programs target women aged 30-49 years, approximately 40% of cervical cancer cases occur after the age of 50. Postmenopausal women face unique anatomical and physiological changes-particularly the regression of the squamocolumnar junction into the endocervical canal-that reduce the sensitivity of visual triage methods such as visual inspection with acetic acid (VIA). Evidence on optimal screening and triage strategies for women aged 50 years and older in LMIC settings is currently lacking.

This feasibility study aims to evaluate the diagnostic performance, acceptability, and clinical outcomes of a cervical cancer screening strategy based on high-risk human papillomavirus (hr-HPV) testing on self-collected vaginal samples, followed by cytology triage of HPV-positive postmenopausal women. The study also explores the added value of extended hr-HPV genotyping to refine risk stratification. The target population includes 500 women aged 50-65 years living in the Mifi Health District, West Cameroon.

At the first visit, eligible women will receive standardized information on cervical cancer and study procedures before providing written informed consent. Participants will then collect a self-obtained vaginal sample, which will be tested onsite using the GeneXpert platform for detection of all hr-HPV types. HPV-negative women will be advised to repeat screening after 5-10 years (or 3-5 years if HIV-positive). HPV-positive women will undergo clinician-collected Pap cytology and endocervical brushing (ECB). Cytology slides will be prepared using manual liquid-based cytology techniques, digitized using a portable whole-slide scanner, and interpreted remotely by trained cytopathologists. ECB samples will undergo histopathological evaluation and will constitute the diagnostic gold standard for assessing triage performance.

Women with cytology results ≥ASC-US will be referred for evaluation and treatment at Bafoussam Regional Hospital. A VIA/VILI examination will guide thermal ablation treatment using WHO-recommended devices and probes adapted to cervical anatomy. Cervical biopsies will be performed in the presence of suspicious lesions suggestive of high-grade disease or cancer. All treatments, follow-up assessments, and management of adverse events will be provided free of charge.

All HPV-positive participants, regardless of baseline cytology results, will be invited for a 12-month follow-up visit including repeat HPV testing, cytology, ECB, and VIA/VILI. Persistence of CIN2+ at 12 months will indicate the need for large loop excision of the transformation zone (LLETZ). Treatment adherence, side effects, and acceptability of the screening and treatment process will be assessed using structured questionnaires administered at baseline, post-treatment (4-6 weeks), and 12 months.

The primary outcomes include sensitivity, specificity, positive and negative predictive values, and likelihood ratios of cytology and extended genotyping (alone or combined) for detection of CIN2+ compared with ECB histology. Secondary outcomes include prevalence of hr-HPV infection and high-grade lesions, effectiveness of thermal ablation for CIN2+ clearance at 12 months, acceptability among women and healthcare providers, and adherence to all steps of the two-stage screening strategy.

This project is expected to generate essential evidence to guide cervical cancer screening policies for older women in LMICs, support the WHO global elimination initiative, and offer a scalable, context-adapted approach combining self-sampling, digital cytology, and appropriate treatment pathways.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 to 65 years old;
* Ability to understand study procedures and accepting voluntarily to participate by signing an informed consent form (ICF).

Exclusion Criteria:

* Women who is pregnant;
* Women with a condition that interfere with visualization of the cervix;
* Women with vaginal bleeding outside the menstrual period;
* Women who have had a total hysterectomy;
* Women with a history of cervical cancer;
* Women screened for cervical cancer in the last 5 years or in the last 3 years if HIV-positive;
* Women in the terminal phase of an illness.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The source population is the entire population of women aged between 50 and 65 years old in the Mifi health district.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of HPV test followed by cytology to detect cervical precancerous lesions in sub-Saharan Africa using histology as gold standard | 1 year
  To determine the diagnostic performance of screening strategies using HPV testing with cytology triage and/or extended genotyping in women aged between 50 and 65 years for the detection of cervical intraepithelial neoplasia grade 2 or worse (CIN2+);

CONTACTS AND LOCATIONS:
Locations (1):
- Bafoussam Regional Hospital, Bafoussam, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided